CLINICAL TRIAL: NCT03159247
Title: The eyeGuide: Improving Glaucoma Self-management With a Personalized Behavior Change Program
Acronym: eyeGuide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Eye Institute (NEI) (NIH); Research to Prevent Blindness (Other); Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Paula Anne Newman-Casey, Assistant Professor of Ophthalmology and Visual Sciences, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00112614; 1K23EY025320-01A1 (NIH)
Record Dates: First submitted 2017-05-12; First posted 2017-05-18 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Medication Adherence; Glaucoma
Keywords: education; counseling; motivational interviewing; tailoring
MeSH Terms: conditions — Medication Adherence; Glaucoma

STUDY DESIGN:
Intervention Model Description: This is a single group prospective behavioral intervention with a pre-post design. Adherence will be measured for three months at baseline, for an additional one month after an automated reminder system is initiated, for an additional six months during a personalized behavior change intervention and then for one year after the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- eyeGuide (Experimental): Two personalized eHealth interventions aimed to improve glaucoma medication adherence.
  Interventions: Behavioral: eyeGuide

INTERVENTIONS:
Behavioral: eyeGuide — The eyeGuide, a web-based tool to facilitate a personalized behavior change program for non-adherent glaucoma patients.

SUMMARY:
The purpose of this research study is to test the impact of two personalized technology based programs that may help improve adherence to glaucoma medications.

DETAILED DESCRIPTION:
Despite evidence from randomized clinical trials that medication reduces vision loss from glaucoma, it remains the second leading cause of blindness in the United States. A critical barrier to preventing vision loss is that about one-half of glaucoma patients are essentially "untreated" because they do not adhere to their medications. Ineffective self-management behaviors and poor clinical outcomes disproportionately affect the most vulnerable members of US society. The increased burden of glaucoma due to an aging US population, together with a projected shortage of ophthalmologists, will make team-based care essential. There is a critical need to develop and test team-based, personalized behavior change interventions for glaucoma patients to improve medication adherence and the outcomes of care.

Poor adherence to effective medications is a critical barrier to better outcomes in glaucoma patients. The World Health Organization stated that "increasing the effectiveness of adherence interventions may have a far greater impact on the health of the population than any improvement in specific medical treatments." Once diagnosed with glaucoma, at least half of patients do not adhere to their glaucoma medication regimen, return for follow-up, or persist with their medications over the longer term. Patients who are not adherent have more severe visual field loss, which leads to steep declines in health-related quality of life and increased risk of falls and motor vehicle accidents.

Adherence to glaucoma medications is rarely addressed during the clinical encounter because education and counseling programs are not part of standard glaucoma care. Focus groups have demonstrated that patients often have a poor understanding of glaucoma and its treatment. In addition to knowledge gaps, patients have numerous concrete and psychological barriers to managing their glaucoma. In addition, eye drop instillation is rarely taught, and many patients cannot properly instill their medications.

Uniform, scripted approaches to improve adherence do not work. However, complex, individualized counseling interventions, especially those based in motivational interviewing (MI), have improved adherence and health outcomes in many chronic diseases. MI is a style of counseling that engages patients by discussing priorities and obstacles to facilitate intrinsic motivation to change health behavior. Few complex interventions based on these successful principles have been rigorously tested and none implemented into glaucoma care. The eyeGuide is a web-based personally tailored behavior change program based on MI principles, a systematic review of the glaucoma adherence literature, and data from focus groups, surveys and iterative beta-testing with glaucoma patients. It provides individually tailored disease information and support to facilitate MI-based conversations between patients and paraprofessional staff to improve medication adherence. Such technology-based electronic health (eHealth) innovations have great potential to extend the reach of physicians by enabling team-based care.

In this pilot study, the study will test the impact of two personalized eHealth technologies on medication adherence among non-adherent glaucoma patients in a pre-post design: 1) real time automated adherence reminders; and 2) the eyeGuide counseling program. The study will explore the effects of these interventions on secondary outcomes including psychosocial mediators of adherence (e.g. motivation, self-efficacy, satisfaction), intraocular pressure (IOP), and IOP fluctuation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of glaucoma, glaucoma suspect or ocular hypertension
* Taking ≥ 1 glaucoma medication
* Age ≥ 40 years
* Non-adherent to glaucoma medications by both self-report and three months of electronic medication monitoring (adherence ≤ 80%)

Exclusion Criteria:

* Cognitive impairment
* Severe mental illness
* Do not administer own glaucoma medications
* Do not speak English

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Electronically monitored glaucoma medication adherence | 22 months
  electronic medication monitoring

SECONDARY OUTCOMES:
Proportion of days covered with medication | 22 months
  monthly pharmacy refill data for glaucoma medications
Change in self-reported medication adherence | 22 months
  Two survey instruments will be used to determine the amount of change in overall adherence
Change in eye drop instillation technique | 4 months elapsed between 4 month and 8 month site visits
  eye drop instillation technique will be video taped and analyzed on the 4 month and 8 month study visits
Change in Intra-ocular Pressure | 22 months
  Intra-ocular pressure will be measured by Goldmann applanation tonometry
Change in Intra-ocular Pressure Fluctuation | 22 months
  Intraocular pressure data will be analyzed to assess a change in pressure fluctuations

CONTACTS AND LOCATIONS:
Overall Officials: Paula A Newman-Casey, MD, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garway-Heath DF, Crabb DP, Bunce C, Lascaratos G, Amalfitano F, Anand N, Azuara-Blanco A, Bourne RR, Broadway DC, Cunliffe IA, Diamond JP, Fraser SG, Ho TA, Martin KR, McNaught AI, Negi A, Patel K, Russell RA, Shah A, Spry PG, Suzuki K, White ET, Wormald RP, Xing W, Zeyen TG. Latanoprost for open-angle glaucoma (UKGTS): a randomised, multicentre, placebo-controlled trial. Lancet. 2015 Apr 4;385(9975):1295-304. doi: 10.1016/S0140-6736(14)62111-5. Epub 2014 Dec 19. PMID 25533656
- [Background] Heijl A, Leske MC, Bengtsson B, Hyman L, Bengtsson B, Hussein M; Early Manifest Glaucoma Trial Group. Reduction of intraocular pressure and glaucoma progression: results from the Early Manifest Glaucoma Trial. Arch Ophthalmol. 2002 Oct;120(10):1268-79. doi: 10.1001/archopht.120.10.1268. PMID 12365904
- [Background] Quigley HA, Broman AT. The number of people with glaucoma worldwide in 2010 and 2020. Br J Ophthalmol. 2006 Mar;90(3):262-7. doi: 10.1136/bjo.2005.081224. PMID 16488940
- [Background] Olthoff CM, Schouten JS, van de Borne BW, Webers CA. Noncompliance with ocular hypotensive treatment in patients with glaucoma or ocular hypertension an evidence-based review. Ophthalmology. 2005 Jun;112(6):953-61. doi: 10.1016/j.ophtha.2004.12.035. PMID 15885795
- [Background] Reardon G, Kotak S, Schwartz GF. Objective assessment of compliance and persistence among patients treated for glaucoma and ocular hypertension: a systematic review. Patient Prefer Adherence. 2011;5:441-63. doi: 10.2147/PPA.S23780. Epub 2011 Sep 23. PMID 22003282
- [Background] Murakami Y, Lee BW, Duncan M, Kao A, Huang JY, Singh K, Lin SC. Racial and ethnic disparities in adherence to glaucoma follow-up visits in a county hospital population. Arch Ophthalmol. 2011 Jul;129(7):872-8. doi: 10.1001/archophthalmol.2011.163. PMID 21746977
- [Background] Congdon N, O'Colmain B, Klaver CC, Klein R, Munoz B, Friedman DS, Kempen J, Taylor HR, Mitchell P; Eye Diseases Prevalence Research Group. Causes and prevalence of visual impairment among adults in the United States. Arch Ophthalmol. 2004 Apr;122(4):477-85. doi: 10.1001/archopht.122.4.477. PMID 15078664
- [Background] Lee PP, Hoskins HD Jr, Parke DW 3rd. Access to care: eye care provider workforce considerations in 2020. Arch Ophthalmol. 2007 Mar;125(3):406-10. doi: 10.1001/archopht.125.3.406. No abstract available. PMID 17353416
- [Background] Sabate E. Adherence to Long-Term Therapies: Evidence for Action. Geneva, Switzerland: World Health Organization (WHO); 2003. Available at: http://www.who.int/chp/knowledge/publications/adherence_full_report.pdf. Accessed June 7, 2015.
- [Background] Kass MA, Gordon M, Morley RE Jr, Meltzer DW, Goldberg JJ. Compliance with topical timolol treatment. Am J Ophthalmol. 1987 Feb 15;103(2):188-93. doi: 10.1016/s0002-9394(14)74225-4. PMID 3812621
- [Background] Newman-Casey PA, Blachley T, Lee PP, Heisler M, Farris KB, Stein JD. Patterns of Glaucoma Medication Adherence over Four Years of Follow-Up. Ophthalmology. 2015 Oct;122(10):2010-21. doi: 10.1016/j.ophtha.2015.06.039. Epub 2015 Aug 25. PMID 26319441
- [Background] Rossi GC, Pasinetti GM, Scudeller L, Radaelli R, Bianchi PE. Do adherence rates and glaucomatous visual field progression correlate? Eur J Ophthalmol. 2011 Jul-Aug;21(4):410-4. doi: 10.5301/EJO.2010.6112. PMID 21140373
- [Background] Sleath B, Blalock S, Covert D, Stone JL, Skinner AC, Muir K, Robin AL. The relationship between glaucoma medication adherence, eye drop technique, and visual field defect severity. Ophthalmology. 2011 Dec;118(12):2398-402. doi: 10.1016/j.ophtha.2011.05.013. PMID 21856009
- [Background] Stewart WC, Chorak RP, Hunt HH, Sethuraman G. Factors associated with visual loss in patients with advanced glaucomatous changes in the optic nerve head. Am J Ophthalmol. 1993 Aug 15;116(2):176-81. doi: 10.1016/s0002-9394(14)71282-6. PMID 8352302
- [Background] McKean-Cowdin R, Varma R, Wu J, Hays RD, Azen SP; Los Angeles Latino Eye Study Group. Severity of visual field loss and health-related quality of life. Am J Ophthalmol. 2007 Jun;143(6):1013-23. doi: 10.1016/j.ajo.2007.02.022. Epub 2007 Apr 2. PMID 17399676
- [Background] McKean-Cowdin R, Wang Y, Wu J, Azen SP, Varma R; Los Angeles Latino Eye Study Group. Impact of visual field loss on health-related quality of life in glaucoma: the Los Angeles Latino Eye Study. Ophthalmology. 2008 Jun;115(6):941-948.e1. doi: 10.1016/j.ophtha.2007.08.037. Epub 2007 Nov 12. PMID 17997485
- [Background] Freeman EE, Munoz B, West SK, Jampel HD, Friedman DS. Glaucoma and quality of life: the Salisbury Eye Evaluation. Ophthalmology. 2008 Feb;115(2):233-8. doi: 10.1016/j.ophtha.2007.04.050. Epub 2007 Jul 26. PMID 17655930
- [Background] Varma R, Wu J, Chong K, Azen SP, Hays RD; Los Angeles Latino Eye Study Group. Impact of severity and bilaterality of visual impairment on health-related quality of life. Ophthalmology. 2006 Oct;113(10):1846-53. doi: 10.1016/j.ophtha.2006.04.028. Epub 2006 Aug 4. PMID 16889831
- [Background] Haymes SA, Leblanc RP, Nicolela MT, Chiasson LA, Chauhan BC. Risk of falls and motor vehicle collisions in glaucoma. Invest Ophthalmol Vis Sci. 2007 Mar;48(3):1149-55. doi: 10.1167/iovs.06-0886. PMID 17325158
- [Background] Sleath B, Blalock SJ, Carpenter DM, Sayner R, Muir KW, Slota C, Lawrence SD, Giangiacomo AL, Hartnett ME, Tudor G, Goldsmith JA, Robin AL. Ophthalmologist-patient communication, self-efficacy, and glaucoma medication adherence. Ophthalmology. 2015 Apr;122(4):748-54. doi: 10.1016/j.ophtha.2014.11.001. Epub 2014 Dec 24. PMID 25542521
- [Background] Sleath BL, Blalock SJ, Muir KW, Carpenter DM, Lawrence SD, Giangiacomo AL, Goldsmith JA, Hartnett ME, Slota C, Robin AL. Determinants of Self-Reported Barriers to Glaucoma Medicine Administration and Adherence: A Multisite Study. Ann Pharmacother. 2014 Jul;48(7):856-862. doi: 10.1177/1060028014529413. Epub 2014 Apr 1. PMID 24692604
- [Background] Lacey J, Cate H, Broadway DC. Barriers to adherence with glaucoma medications: a qualitative research study. Eye (Lond). 2009 Apr;23(4):924-32. doi: 10.1038/eye.2008.103. Epub 2008 Apr 25. PMID 18437182
- [Background] Stryker JE, Beck AD, Primo SA, Echt KV, Bundy L, Pretorius GC, Glanz K. An exploratory study of factors influencing glaucoma treatment adherence. J Glaucoma. 2010 Jan;19(1):66-72. doi: 10.1097/IJG.0b013e31819c4679. PMID 20075676
- [Background] Taylor SA, Galbraith SM, Mills RP. Causes of non-compliance with drug regimens in glaucoma patients: a qualitative study. J Ocul Pharmacol Ther. 2002 Oct;18(5):401-9. doi: 10.1089/10807680260362687. PMID 12419091
- [Background] Lunnela J, Kaariainen M, Kyngas H. The views of compliant glaucoma patients on counselling and social support. Scand J Caring Sci. 2010 Sep;24(3):490-8. doi: 10.1111/j.1471-6712.2009.00739.x. PMID 20210901
- [Background] Newman-Casey PA, Robin AL, Blachley T, Farris K, Heisler M, Resnicow K, Lee PP. The Most Common Barriers to Glaucoma Medication Adherence: A Cross-Sectional Survey. Ophthalmology. 2015 Jul;122(7):1308-16. doi: 10.1016/j.ophtha.2015.03.026. Epub 2015 Apr 24. PMID 25912144
- [Background] Friedman DS, Hahn SR, Gelb L, Tan J, Shah SN, Kim EE, Zimmerman TJ, Quigley HA. Doctor-patient communication, health-related beliefs, and adherence in glaucoma results from the Glaucoma Adherence and Persistency Study. Ophthalmology. 2008 Aug;115(8):1320-7, 1327.e1-3. doi: 10.1016/j.ophtha.2007.11.023. Epub 2008 Mar 5. PMID 18321582
- [Background] Tsai JC, McClure CA, Ramos SE, Schlundt DG, Pichert JW. Compliance barriers in glaucoma: a systematic classification. J Glaucoma. 2003 Oct;12(5):393-8. doi: 10.1097/00061198-200310000-00001. PMID 14520147
- [Background] Hennessy AL, Katz J, Covert D, Kelly CA, Suan EP, Speicher MA, Sund NJ, Robin AL. A video study of drop instillation in both glaucoma and retina patients with visual impairment. Am J Ophthalmol. 2011 Dec;152(6):982-8. doi: 10.1016/j.ajo.2011.05.015. Epub 2011 Aug 6. PMID 21821228
- [Background] Sleath B, Blalock SJ, Stone JL, Skinner AC, Covert D, Muir K, Robin AL. Validation of a short version of the glaucoma medication self-efficacy questionnaire. Br J Ophthalmol. 2012 Feb;96(2):258-62. doi: 10.1136/bjo.2010.199851. Epub 2011 May 24. PMID 21610264
- [Background] Waterman H, Evans JR, Gray TA, Henson D, Harper R. Interventions for improving adherence to ocular hypotensive therapy. Cochrane Database Syst Rev. 2013 Apr 30;2013(4):CD006132. doi: 10.1002/14651858.CD006132.pub3. PMID 23633333
- [Background] Nieuwlaat R, Wilczynski N, Navarro T, Hobson N, Jeffery R, Keepanasseril A, Agoritsas T, Mistry N, Iorio A, Jack S, Sivaramalingam B, Iserman E, Mustafa RA, Jedraszewski D, Cotoi C, Haynes RB. Interventions for enhancing medication adherence. Cochrane Database Syst Rev. 2014 Nov 20;2014(11):CD000011. doi: 10.1002/14651858.CD000011.pub4. PMID 25412402
- [Background] Newman-Casey PA, Weizer JS, Heisler M, Lee PP, Stein JD. Systematic review of educational interventions to improve glaucoma medication adherence. Semin Ophthalmol. 2013 May;28(3):191-201. doi: 10.3109/08820538.2013.771198. PMID 23697623
- [Background] Newman-Casey PA, Shtein RM, Coleman AL, Herndon L, Lee PP. Why Patients With Glaucoma Lose Vision: The Patient Perspective. J Glaucoma. 2016 Jul;25(7):e668-75. doi: 10.1097/IJG.0000000000000320. PMID 26317482
- [Background] Miller WR and Rollnick S. Motivational Interviewing: Helping people change, 3rd edition. 2013; Guilford Press, New York, NY.
- [Derived] Schneider KJ, Hollenhorst CN, Valicevic AN, Niziol LM, Heisler M, Musch DC, Cain SM, Newman-Casey PA. Impact of the Support, Educate, Empower Personalized Glaucoma Coaching Program Pilot Study on Eye Drop Instillation Technique and Self-Efficacy. Ophthalmol Glaucoma. 2021 Jan-Feb;4(1):42-50. doi: 10.1016/j.ogla.2020.08.003. Epub 2020 Aug 8. PMID 32781286
- [Derived] Sanchez FG, Mansberger SL, Newman-Casey PA. Predicting Adherence With the Glaucoma Treatment Compliance Assessment Tool. J Glaucoma. 2020 Nov;29(11):1017-1024. doi: 10.1097/IJG.0000000000001616. PMID 32740508
- [Derived] Newman-Casey PA, Niziol LM, Mackenzie CK, Resnicow K, Lee PP, Musch DC, Heisler M. Personalized behavior change program for glaucoma patients with poor adherence: a pilot interventional cohort study with a pre-post design. Pilot Feasibility Stud. 2018 Jul 23;4:128. doi: 10.1186/s40814-018-0320-6. eCollection 2018. PMID 30062043